CLINICAL TRIAL: NCT02141256
Title: Can Protein Intake be Increased by Offering Protein-enriched Foods and Drinks? Evaluation of a Pilot in a Local Residential Care Home.
Brief Title: Can Protein Intake be Increased by Offering Protein-enriched Foods and Drinks?
Acronym: EET-studie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL45883.081.13
Record Dates: First submitted 2013-10-29; First posted 2014-05-19 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Undernutrition
Keywords: elderly; protein enrichment; undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Protein enriched products (Experimental): Protein enriched products will be given to elderly residents of a care home for 10 days. Does this lead to an increased protein intake or do elderly compensate for the extra amount of protein?
  Interventions: Dietary Supplement: Protein enriched products

INTERVENTIONS:
Dietary Supplement: Protein enriched products — Newly developed products with extra protein. Specially developed for elderly.

SUMMARY:
The objective of this study is to investigate whether a protein-enriched daily menu is acceptable and effective in increasing protein intake in elderly in a residential care home up to an intake of 1,2 gram/ kg body weight per day.

The investigators hypothesise that when elderly eat 2 slices of bread, 1 portion of juice and 1 portion of soup each day, the protein intake can be increased by at least 20 grams/day. On average this can lead to an intake of 1,2 gram/ kg body weight per day.

DETAILED DESCRIPTION:
Rationale: Due to inactivity, elderly are prone to lose muscle mass. With an increased protein intake, muscle mass might be maintained. The current recommendation for protein intake for elderly is the same as for younger adults, but researchers and geriatricians appeal for a higher recommended protein intake to maintain health and function. One way to reach a higher intake is by providing protein-enriched foods. Because of concerns that these foods are more satiating, careful monitoring of protein intake after introducing these foods is warranted.

Objective: To investigate whether a protein-enriched daily menu is acceptable and effective in increasing protein intake in elderly in a residential care home up to an intake of 1,2 gram/ kg body weight per day.

Study design: Dietary intake will be monitored before and after introducing a protein-enriched daily menu. The menu will be provided for 10 days to all residents of the care home. For residents who give consent, intake will be recorded by trained research assistants and nurses on 2 consecutive days before the pilot and on days 9 and 10 of the pilot. After the pilot residents will return to their regular menus.

Study population: The study population consists of elderly men and women (aged 65 or older) living in a care home in Wageningen, the Netherlands.

Intervention: A protein-enriched daily menu for 10 days.

Main study parameters/endpoints: Protein intake and resident satisfaction with the menu.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* living in care home Nudehof
* able to give consent
* without dietary protein restrictions

Exclusion Criteria:

* cognitive impaired
* having dementia
* having dysphagia
* receiving only tube feeding
* known kidney disease
* having food allergies that exclude them from having the protein-enriched products
* following a low protein diet or a diet low in sodium
* receiving palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in protein intake | baseline, day 9 and 10 of intervention

SECONDARY OUTCOMES:
Satisfaction with newly developed products | all days of intervention participants will be followed, an average of 10 days
  Qualitative measurement

CONTACTS AND LOCATIONS:
Overall Officials: N M de Roos, PhD, Principal Investigator — Wageningen University
Locations (1):
- Nudehof, Wageningen, Gelderland, Netherlands